CLINICAL TRIAL: NCT05647850
Title: Optimization and Clinical Study of Early Prediction Model for Neonatal Acute Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University-Town Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hui Liu, Attending physician, University-Town Hospital of Chongqing Medical University
Other Study IDs: 123456
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Neonatology
Keywords: Neonatal acute respiratory distress syndrome; Model of prediction; Perinatal factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Umbilical cord blood was used to test inflammatory markers of Umbilical cord blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline characteristics of all patients
  Interventions: Other: No intervention
- General characteristics of the patients.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this observational study is to learn about neonatal acute respiratory distress syndrome in describe participant population. The main question it aims to answer is: using perinatal factors to predict early neonatal acute respiratory distress syndrome and reduce its mortality.

Participants' umbilical cord blood will be collected for testing, but will not receive any intervention.

ELIGIBILITY:
Inclusion Criteria:

* A newborn born alive

Exclusion Criteria:

* Stillborn newborn
* Respiratory distress syndrome(RDS), transient tachypnoea of the neonate (TTN), or congenital anomalies as a primary current acute respiratory condition
* Hereditary endocrine and metabolic diseases
* Incomplete records

Min Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All infants from a multi-center study in China, will hospitalise between January 1, 2023 and December 31, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
General characteristics of the patients | 2023.1-2025.12

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Principal Investigator — University-Town Hospital of Chongqing Medical University
Locations (2):
- China (2):
  - University-Town Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Women and Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No